CLINICAL TRIAL: NCT00527293
Title: Partial Breast Irradiation for Patients Undergoing Breast Conservation Therapy for Early Stage Breast Cancer: A Pilot Study
Brief Title: Partial Breast Radiation Therapy in Treating Women Undergoing Breast-Conserving Therapy for Early Stage Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2104; P30CA043703 (NIH); CASE2104 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; invasive ductal breast carcinoma; medullary ductal breast carcinoma with lymphocytic infiltrate; mucinous ductal breast carcinoma; tubular ductal breast carcinoma; papillary ductal breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast | interventions — Chemotherapy, Adjuvant; Radiotherapy, Conformal; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MammoSite Brachytherapy (Experimental): Patients undergo partial breast irradiation comprising either MammoSite® brachytherapy twice daily for 5-10 days
  Interventions: Procedure: adjuvant therapy; Radiation: brachytherapy
- 3-dimensional conformal radiotherapy (Experimental): 3-dimensional conformal radiotherapy twice daily for 5-10 days.
  Interventions: Procedure: adjuvant therapy; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Procedure: adjuvant therapy — If chemotherapy is planned, it must begin no earlier than two weeks following completion of radiation. If chemotherapy is given first, a minimum of 2 weeks from the last cycle must elapse prior to the start of radiation.
Radiation: 3-dimensional conformal radiation therapy — 3-dimensional conformal radiotherapy twice daily for 5-10 days.
  Arms: 3-dimensional conformal radiotherapy
Radiation: brachytherapy — Patients undergo partial breast irradiation comprising either MammoSite® brachytherapy twice daily for 5-10 days
  Arms: MammoSite Brachytherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Giving radiation therapy in different ways may kill more tumor cells.

PURPOSE: This clinical trial is studying how well partial breast radiation therapy works in treating women undergoing breast-conserving therapy for early stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the cosmetic outcome resulting from partial breast irradiation using two different techniques.
* To determine patient satisfaction with partial breast irradiation as it pertains to their overall treatment experience as measured by a questionnaire.
* To determine if there are patient factors that limit a patient's suitability to receive partial breast irradiation delivered by a particular technique.
* To evaluate wound healing and overall complication rate after partial breast irradiation.
* To determine ipsilateral breast tumor recurrence rates and tumor bed recurrence rates.

OUTLINE: Patients undergo partial breast irradiation comprising either MammoSite® brachytherapy twice daily for 5-10 days OR 3-dimensional conformal radiotherapy twice daily for 5-10 days.

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer, including the following histologic subtypes:

  * Invasive ductal carcinoma
  * Medullary ductal carcinoma
  * Papillary ductal carcinoma
  * Colloid (mucinous) ductal carcinoma
  * Tubular ductal carcinoma
* The following histologic subtypes are not allowed:

  * Invasive lobular carcinoma
  * Extensive lobular carcinoma in situ
  * Ductal carcinoma in situ (DCIS)
  * Nonepithelial breast malignancies, such as lymphoma or sarcoma
* No extensive intraductal component by Harvard definition (i.e., more than 25% of the invasive tumor is DCIS or DCIS present in adjacent tissue)
* Stage I or II disease (T1, N0; T1, N1a; T2, N0; or T2, N1a)

  * Lesion ≤ 3 cm
  * No more than 3 positive lymph nodes

    * Patients with 4 or more positive axillary lymph nodes found at the time of axillary lymph node dissection/sentinel lymph node biopsy are not eligible
* Has undergone tylectomy (lumpectomy) and axillary lymph node sampling (axillary node dissection or sentinel node biopsy)

  * Negative resection margins with ≥ 2 mm margin from invasive or in situ cancer OR a negative re-excision margin
* Unifocal breast cancer

  * No multicentric carcinoma (tumors in different quadrants of the breast or tumors separated by ≥ 4 cm)

    * No palpable or radiographically suspicious contralateral axillary, ipsilateral or contralateral supraclavicular, infraclavicular, or internal mammary lymph nodes unless these are histologically confirmed negative
* No skin involvement of disease
* No Paget's disease of the nipple
* No distant metastatic disease
* Hormone-receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Not pregnant or lactating
* Negative pregnancy test
* Fertile patients must use effective contraception for ≥ 1 week prior to, during, and for ≥ 2 weeks after completion of study treatment
* No collagen vascular disorders, specifically systemic lupus erythematosus, scleroderma, or dermatomyositis
* No psychiatric, neurologic, or addictive disorders that would preclude obtaining informed consent
* No other malignancy within the past 5 years, except non-melanomatous skin cancer

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the breast
* No chemotherapy for at least 2 weeks before and 2 weeks after completion of study radiotherapy
* Concurrent hormonal therapy allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-06; Primary Completion 2010-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Cosmetic outcome as determined by an established scale employed by the radiation oncologist and the surgeon | 1 month after RT & Q3mos for one year
Patient satisfaction with partial breast irradiation as measured by a questionnaire | Pre-treatment 1 mo 3 mo 6 mo 9 mo 1yr 5 yr
Wound healing and overall complication rate after partial breast irradiation | 1 month after RT & Q3mos for one year
Determination of which patients are best suited for each individual technique of partial breast irradiation | Patients will be followed for a period of five years following completion of radiation.
Ipsilateral breast tumor recurrence rates and tumor bed recurrence rates | Ipsilateral breast 6 mos after dx, bilateral annually x 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Janice Lyons, MD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Lake/University Ireland Cancer Center, Cleveland, Ohio
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio